CLINICAL TRIAL: NCT03673644
Title: Glaucoma, Visual Field Loss, and Their Association With Life Space in Older Adults
Brief Title: Impact of Glaucoma and Visual Field Loss on Life Space
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lyne Racette, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300001552; 5P30AG022838-14 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary Open-Angle Glaucoma: Two following two questionnaires will be administered:
  1. Life Space Questionnaire: This 9-item questionnaire is interested in finding out how much a person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame.
  2. Low Luminance Questionnaire: This 32-item questionnaire is interested in finding out problems that involve vision under different lighting conditions or feelings that people have about your vision under different lighting conditions.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Two questionnaires will be administered, one focusing on life space and the other focusing on low luminance.

SUMMARY:
Mobility refers to a person's purposeful movement through the environment from one place to another and can be conceptualized as a continuum from bed bound (immobility) on one extreme to making excursions to distant locations on the other extreme. Primary open-angle glaucoma (POAG) is a chronic, progressive optic neuropathy that can lead to gradual loss of vision in the peripheral field and central vision. Older adults with POAG have an increased risk for motor vehicle collisions and falls. Moreover, existing studies suggest that patients with POAG exhibit more postural sway while standing as measured by a balance platform and also tend to walk more slowly than those who are normally sighted and free of ocular disease. While these disturbances likely influence mobility, there has been little research directly assessing the impact of POAG on mobility. This study will assess the impact of POAG on life space (one aspect of mobility) and will determine whether difficulties with life space are associated with difficulties experienced under conditions of dim lighting.

DETAILED DESCRIPTION:
Aim 1: To examine the extent of life space in older adults with POAG using the Life Space Questionnaire and to examine whether life space in persons with POAG is associated with the magnitude of visual field impairment.

Aim 2: To examine difficulties seeing under dim illumination and at night in older adults with POAG using the Low Luminance Questionnaire and to examine whether greater difficulty in seeing under dim illumination and at night is related to the magnitude of visual field loss.

Aim 3: To examine the relationship in older adults with POAG between visual problems seeing under dim illumination and at night (Low Luminance Questionnaire) and their life space (Life Space Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary open-angle glaucoma
* Best-corrected visual acuity of 20/40 or better
* Spherical refraction within ± 5 Diopters
* Cylinder refraction within ± 3 Diopters

Exclusion Criteria:

* History of intra-ocular surgery other than uncomplicated cataract or glaucoma surgery
* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that are enrolled in the Early Detection of Glaucoma Progression using a Novel Individualized Approach (IRB-300000301) or in the African Descent and Glaucoma Evaluation (ADAGES) IV: Alterations of the Lamina Cribrosa in Progression (IRB-161115004).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of life space measured with the Life Space Questionnaire | Day one
  The Life Space Questionnaire is a 9-item questionnaire that assesses how much a person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame. Patients are asked to respond either Yes or No.

SECONDARY OUTCOMES:
Relationship between the Life Space Questionnaire and vision loss | Day one
  The results obtained on the Life Space Questionnaire will be correlated with the results of the visual field tests
Assessment of vision under dim illumination and at night using the Low Luminance Questionnaire | Day one
  The Low Luminance Questionnaire is a 32-item questionnaire that assesses problems that involve vision under different lighting conditions or feelings about vision under different lighting conditions. The range of responses is different for different questions, with the overall pattern being that "1" means "No difficulty at all" and that increasingly higher numbers mean increasingly more difficulty.
Relationship between Low Luminance Questionnaire and vision loss | Day one
  The results obtained on the Low Luminance Questionnaire will be correlated with the results of the visual field tests.
Relationship between the Low Luminance Questionnaire and the Life Space Questionnaire | Day one
  The results of the Low Luminance Questionnaire will be correlated with the results of the Life Space Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lyne Racette, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share our redacted individual participant data with other researchers at the time of sharing results.